CLINICAL TRIAL: NCT04102800
Title: Asthma Exacerbation Profile in Patients on Open Label Treatment With Benralizumab for Severe Eosinophilic Asthma - an Exploratory Cohort Study
Brief Title: Benralizumab Exacerbation Study
Acronym: BenRex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); AstraZeneca (Industry); Queen's University, Belfast (Other); Bosch Healthcare Solutions GmbH (Industry); InHealthcare (Unknown); University of Leicester (Other); University of Plymouth (Other); Vitalograph (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN17RM684
Record Dates: First submitted 2019-03-12; First posted 2019-09-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: benralizumab; exacerbation; eosinophilic
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Benralizumab 30mg by subcutaneous injection, 18 months treatment for the first 75 participants enrolled, 12 months treatment for participants 76-150
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — subcutaneous injection

SUMMARY:
This is an exploratory study, the focus of which is to understand the nature of asthma exacerbations that occur despite open label benralizumab therapy in severe eosinophilic asthma.

DETAILED DESCRIPTION:
A phase IV, open-label, prospective, multi-centre cohort study in patients with severe eosinophilic asthma (Global Initiative for Asthma [GINA] steps 4 and 5 classification of asthma severity) who will be treated with benralizumab injections. The study is exploratory and will assess deteriorations in asthma control (exacerbations) to characterise the clinical severity of each exacerbation and the airway and systemic inflammatory phenotype associated with these events. Clinical assessment and management of each exacerbation will be in line with standard clinical guidelines. 150 participants will be recruited and receive treatment for either 56 or 80 weeks.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to provide written informed consent and to comply with the study protocol, including being able to attend for assessment during a symptomatic deterioration
* severe asthma confirmed after assessment by an asthma specialist, requiring treatment with high dose inhaled corticosteroids (ICS) as per BTS criteria [>1000 fluticasone proportionate equivalent] and >1 additional drug for asthma (e.g. long acting beta 2 antagonist (LABA)/leukotriene receptor antagonist/theophylline/long acting muscarinic antagonist) at screening [participants may be included with a lower dose of current ICS at the discretion of the investigator if previous high ICS dose had led to side effects]
* Adherent with background asthma medication in the opinion of the investigator [adherence assessments as per local practice]
* Assessed and treatment optimised for any significant asthma-related co-morbidities
* Considered suitable by an asthma specialist for treatment with a monoclonal antibody to block the Interleukin-5 pathway as per local practice. Participants will have: a) recorded blood eosinophil count ≥0.3 x 109/L within the past year along with a history of either ≥4 asthma exacerbations requiring high dose oral corticosteroids* and/or maintenance systemic corticosteroids equivalent to prednisolone ≥5 mg/day for 6 months or longer OR b) recorded blood eosinophil count ≥0.4 x 109/L within the past year along with a history of ≥ 3 asthma exacerbations requiring high dose oral corticosteroids*

  * [Exacerbations of asthma in the past year will be defined as worsening of asthma symptoms leading to treatment with prednisolone ≥30 mg oral corticosteroids for ≥3 days or an increase ≥ 10mg in oral corticosteroids for at least 3 days for patients on maintenance oral steroids] as defined by the ERS/ATS Task Force

Exclusion Criteria:

* Acute exacerbation requiring high dose oral corticosteroids in the 2 weeks prior to Visit 1 or during the screening period. Such patients would be re-assessed after 2 weeks for re-screening.
* Other clinically significant medical disease or uncontrolled concomitant disease that is likely, in the opinion of the investigator, to require a change in therapy or impact the ability to participate in the study.
* History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the subject's full participation in the study, in the opinion of the investigator.
* Female patients who are pregnant or lactating or planning a family
* Active lung disease other than asthma [Note: Controlled obstructive sleep apnoea (OSA), minor bronchiectasis, asbestos pleural plaques or old (inactive) TB scars are not exclusion criteria]. Patients where an asthma-COPD overlap is suspected by the investigator are not eligible for inclusion.
* Current smoker [history of smoking [including e-cigarettes] in the past 3 months prior to Visit 1.
* Treatment with any of the following prior to Visit 1 or during the study

  1. any biologic medicine for asthma or an immunomodulating biologic agent for other conditions in the 3 months prior to Visit 1
  2. an investigational agent within 30 days of Visit 1 (or five half lives of the investigational agent, whichever is longer).
  3. Administration of live attenuated vaccine 30 days prior to Visit 1. Other types of approved vaccines are allowed.
  4. Regular use of systemic (oral/IM) corticosteroids except for the indication of asthma or adrenal insufficiency [note: patients taking systemic steroid replacement primarily for adrenal insufficiency can be included provided they meet exacerbation inclusion criteria]
  5. Other ongoing immunosuppressive/ immunomodulating therapy [e.g. methotrexate, ciclosporine, azathioprine] other than oral corticosteroids for asthma.
* Bronchial thermoplasty conducted within 6 months of Visit 1.
* History of known immunodeficiency disorder including a previous positive human immunodeficiency virus (HIV) test
* Active or suspected Helminth infection. Patients with helminth infections must be excluded until the infection has been treated
* Known hypersensitivity to benralizumab (the active substance) or any of the excipients [Histidine, Histidine hydrochloride monohydrate, Trehalose dihydrate, Polysorbate 20, water for injections]
* Women of child bearing potential (WoCBP) who are not willing to use highly effective contraception during treatment with benralizumab and for 16 weeks after the last dose. WoCBP will be required to undergo a urine pregnancy test prior to administration of each benralizumab injection.
* Current malignancy, or history of malignancy, except for:

  1. patients who have had non-melanoma skin cancers or in situ carcinoma of the cervix - these patients are eligible provided that the patient is in remission and curative therapy was completed at least 12 months prior to the date informed consent is obtained. b) Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to the date informed consent is obtained.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Blood eosinophil counts during a clinical deterioration whilst on benralizumab | up to 56 or 80 weeks
Fall in lung function, as measured by FEV1, during a clinical deterioration whilst on benralizumab. | up to 56 or 80 weeks
Change in asthma symptom scores during a clinical deterioration whilst on benralizumab. | up to 56 or 80 weeks
The number of patients progressing to rescue oral corticosteroids during a clinical deterioration whilst on benralizumab. | up to 56 or 80 weeks

SECONDARY OUTCOMES:
Measurement of the magnitude of response to benralizumab - oral steroid reduction with benralizumab at 56 weeks | 56 weeks
  proportion of patients who reduce high dose steroid courses and/or maintenance steroid dose by >=25%, 50%, 75% and 100%
Measurement of the magnitude of response to benralizumab - numbers of participants with and early and final good response | 16, 24 weeks, 1 year
  Early (16/24 weeks): A GETE response of 'good' or 'excellent' to treatment with benralizumab as determined by the study physician. Final (one year): defined as a reduction of high dose corticosteroid courses by >=50% compared to the previous year and/or reduction of maintenance oral steroid dose by >=50%
Measurement of the magnitude of response to benralizumab - inflammatory markers at 16 and 56 weeks compared to baseline | 16, 56 weeks
  FBC to include Blood eosinophils, sputum eosinophils, blood neutrophil counts
Measurement of the magnitude of response to benralizumab - inflammatory markers at 16 and 56 weeks compared to baseline | 16, 56 weeks
  Measurement of exhaled nitric oxide
Measurement of the magnitude of response to benralizumab - change in lung function, as measured by FEV1, at 16, 24 and 56 weeks compared to baseline | 16, 24 and 56 weeks
  FEV1 post salbutamol on spirometry and FEV1 in daily diary
Measurement of the magnitude of response to benralizumab - change in lung function at 16, 24 and 56 weeks compared to baseline | 16, 24 and 56 weeks
  peak expiratory flow from the daily electronic meter
Measurement of the magnitude of response to benralizumab - change in patient reported outcomes at 16,24 and 56 weeks compared to baseline | 16, 24 and 56 weeks
  Completion of health outcome questionnaires
Identifying predictors of treatment response | 16 weeks and 1 year
  Patients will be classified into treatment responders and non-responders. Logistic regression will be used to identify the predictive value of improvement in early clinical response indicators at 16 weeks on 12 month treatment response.
Comparing patient reported outcome measures | 16, 24 and 56 weeks
  Correlation of completed questionnaires: Scores, and changes in scores, from the SAQ will be correlated with the SGRQ and mini-AQLQ. The SAQ score will be evaluated against demographic features at baseline.
Onset of clinical response | up to 56 or 80 weeks
  Time to first exacerbation and change in FEV1 with time.
Exploratory Microbiomics | baseline, 4, 16 and 56 weeks, during exacerbation visits
  Samples will be stored for later laboratory biomarker measurements. To assess possible biomarkers of response
Exploratory viromics | baseline, 4, 16 and 56 weeks, during exacerbation visits
  Samples will be stored for later laboratory biomarker measurements. To assess possible biomarkers of response
Exploratory transcriptomics | baseline, 4, 16 and 56 weeks, during exacerbation visits
  Samples will be stored for later laboratory biomarker measurements. To assess possible biomarkers of response
Exploratory biomarkers related to asthmatic airway inflammation, corticosteroid signalling and putative inflammatory pathways | baseline, 4, 16 and 56 weeks, during exacerbation visits
  Samples will be stored for later laboratory biomarker measurements. To assess possible biomarkers of response

OTHER OUTCOMES:
Validation of home spirometry with video supported tests | Baseline, 2 and 24 weeks
  Comparison of spirometry done on site with another done off site with video support from the study team.

CONTACTS AND LOCATIONS:
Locations (15):
- United Kingdom (15):
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Gartnavel General Hospital, Glasgow
  - Castle Hill Hospital, Hull
  - Glenfield Hospital, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Guy's and St Thomas's Hospital, London
  - Royal Brompton Hospital, London
  - Royal Free Hospital, London
  - Wythenshawe Hospital, Manchester
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - Queen Alexandra Hospital, Portsmouth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butler CA, Heaney LG. Fractional exhaled nitric oxide and asthma treatment adherence. Curr Opin Allergy Clin Immunol. 2021 Feb 1;21(1):59-64. doi: 10.1097/ACI.0000000000000704. PMID 33369570